CLINICAL TRIAL: NCT02834793
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Trial With an Open-Label Extension Phase of Perampanel as Adjunctive Treatment in Subjects at Least 2 Years of Age With Inadequately Controlled Seizures Associated With Lennox-Gastaut Syndrome
Brief Title: Study of Perampanel as Adjunctive Treatment for Inadequately Controlled Seizures Associated With Lennox-Gastaut Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2007-G000-338; 2014-002321-35 (EudraCT Number)
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2021-03

CONDITIONS: Lennox-Gastaut Syndrome (LGS)
Keywords: Lennox-Gastaut Syndrome (LGS); Inadequately controlled seizures
MeSH Terms: conditions — Lennox Gastaut Syndrome | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Perampanel up to 8 mg/day (Experimental): During the Randomization Phase, participants will receive perampanel at a starting dose of 2 milligrams per day (mg/day). Thereafter, the dose will be increased to a maximum target dose of 8 mg/day according to individual tolerability and efficacy for up to 18 weeks. Participants who enter into Extension A will continue to receive perampanel at the dose last received during randomization phase. Participants can be titrated up to 12 mg/day (at 2-week intervals) per the investigator's discretion.
  Participants who continue in Extension B will continue to receive perampanel at the dose last received at the end of Extension A.
  Interventions: Drug: Perampanel
- Matching placebo (Placebo Comparator): During the Randomization Phase, participants will receive matching placebo for up to 18 weeks.
  During the Extension A, participants who received placebo during the Randomization Phase will begin treatment with perampanel in a blinded manner in double-blind Conversion Period, starting at 2 mg/day and then up-titrated to a maximum target dose of 8 mg/day according to individual tolerability and efficacy. After the Conversion Period, participants can be titrated up to 12 mg/day (at 2-week intervals) per the investigator's discretion.
  Interventions: Drug: Placebo; Drug: Perampanel

INTERVENTIONS:
Drug: Placebo — Participants will receive matching placebo in Randomization phase.
  Arms: Matching placebo
Drug: Perampanel — Participants will receive perampanel in Randomization phase, open-label Extension A, and open-label Extension B.
  Other Names: E2007

SUMMARY:
This study is being conducted to demonstrate that perampanel given as adjunctive anti-epileptic treatment is superior to placebo in reducing the number of drop seizures in participants with inadequately controlled seizures associated with Lennox-Gastaut Syndrome (LGS).

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, placebo-controlled, parallel-group study of perampanel as adjunctive therapy in participants with inadequately controlled seizures associated with LGS. The study will consist of 3 phases: Prerandomization (4 to 8 weeks), Randomization (18 weeks), and an Extension A (52 weeks). An additional Extension B with open-label treatment will be available for optional participation to participants who reside in Japan and in countries where an expanded access program (EAP) cannot be implemented or has not yet been implemented.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of LGS as evidenced by:

  1. more than one type of generalized seizure, including drop seizures (atonic, tonic, or myoclonic) for at least 6 months before Visit 1;
  2. an electroencephalogram (EEG) reporting diagnostic criteria for LGS at some point in their history (abnormal background activity accompanied by slow, spike, and wave pattern <2.5 hertz [Hz]).
* Participants must be at least 2 years old at the time of consent/assent
* Participants must have been <11 years old at the onset of LGS
* Participants must have experienced an average of at least 2 drop seizures per week in the 4-week Baseline Period preceding randomization
* Participants must have been receiving 1 to 4 concomitant antiepileptic drugs (AEDs) at a stable dose for at least 30 days before Visit 1 (vagal nerve stimulation (VNS) and ketogenic diet do not count as AEDs). Use of cannabidiol (CBD) products is allowed and is counted as one of the 4 maximum allowed concomitant AEDs. CBD dose and product must have remained stable for at least 30 days before Visit 1 and is to remain the same throughout the course of the Core Study
* In the investigator's opinion, parents or caregivers must be able to keep accurate seizure diaries
* Body weight at least 8 kilogram (kg)

Exclusion Criteria:

* Presence of progressive neurological disease
* Presence of drop seizure clusters where individual seizures cannot be reliably counted (seizure clusters are defined as ≥2 drop seizures with <5 minutes between any 2 consecutive seizures)
* Prior treatment with perampanel with discontinuation due to safety issues (related to perampanel)
* Prior treatment with perampanel within 30 days before Visit 1
* Evidence of clinically significant disease (eg, cardiac, respiratory, gastrointestinal, renal disease, hepatic disease) that in the opinion of the investigator(s) could affect the participant's safety or study conduct
* Scheduled for epilepsy-related surgery or any other form of surgery during the projected course of the study
* Ketogenic diet and VNS, unless stable and ongoing for at least 30 days before Visit 1
* Treatment with an investigational drug or device within 30 days before Visit 1
* Status epilepticus within 12 weeks of Visit 1
* If felbamate is used as a concomitant AED, participants must be on felbamate for at least 1 year, with a stable dose for 60 days before Visit 1. They must not have a history of white blood cell (WBC) count below ≤2500/microliters (μL), platelets <100,000/μL, liver function tests (LFTs) >3 times the upper limit of normal (ULN), or other indication of hepatic or bone marrow dysfunction while receiving felbamate
* Concomitant use of vigabatrin: participants who took vigabatrin in the past must be discontinued for at least 5 months before Visit 1, and must have documentation showing no evidence of a vigabatrin-associated clinically significant abnormality in an automated visual perimetry test
* Have had multiple drug allergies or a severe drug reaction to an AED(s), including dermatological (eg, Stevens-Johnson syndrome), hematological, or organ toxicity reactions
* Evidence of significant active hepatic disease. Stable elevations of liver enzymes, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) due to concomitant medication(s) will be allowed if they are < 3 times the ULN
* Adrenocorticotropic hormone within the 6 months before Visit 1
* Had history of anoxic episodes requiring resuscitation within 6 months before Visit 1
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta human chorionic gonadotropin [ß-hCG] with a minimum sensitivity of 25 International Units per Liter (IU/L) or equivalent units of ß-hCG or hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
* Females of childbearing potential who: a. had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period or for 28 days after study drug discontinuation. Females using hormonal contraceptives containing levogesterol must be on another form of contraception as well. b. Are currently abstinent, and do not agree to use a double-barrier method (as described above) or refrain from sexual activity during the study period or for 28 days after study drug discontinuation. c. Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study or for 28 days after study drug discontinuation. (NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal [amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause] or have been sterilized surgically [i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing])
* Had intermittent use of benzodiazepine of more than 4 single administrations in the month before Visit 1
* A prolonged QT/QTc interval (QTc >450 milliseconds [ms]) as demonstrated by a repeated electrocardiogram (ECG)
* Hypersensitivity to the study drug or any of the excipients
* Any history of a medical condition or a concomitant medical condition that in the opinion of the investigator(s) would compromise the participant's ability to safely complete the study
* Known to be human immunodeficiency virus (HIV) positive
* Active viral hepatitis (B or C) as demonstrated by positive serology at Screening
* Psychotic disorder(s) or unstable recurrent affective disorder(s) evident by use of antipsychotics or prior suicide attempt(s) within approximately the last 2 years
* History of drug or alcohol dependency or abuse within approximately the last 2 years; use of illegal recreational drugs
* Concomitant use of medications known to be inducers of cytochrome P450 (CYP3A) including, but not limited to: rifampin, troglitazone, St. John's Wort, efavirenz, nevirapine, glucocorticoids (other than topical usage), modafinil, pioglitazone, and rifabutin
* Use of AEDs not recommended by Epilepsy Treatment Guidelines for use in LGS including, but not limited to carbamazepine, gabapentin, oxcarbazepine, phenytoin, pregabalin, tiagabine, and vigabatrin
* Any suicidal ideation with intent with or without a plan within 6 months before Visit 2 (that is, answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the Columbia Suicide Severity Rating Scale (C -SSRS) in participants aged 8 and above.
* Participants with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (31):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford University, Palo Alto, California
  - Northwest Florida Clinical Research Group, LLC, Gulf Breeze, Florida
  - University of Florida Jacksonville, Jacksonville, Florida
  - Pediatric Neurologists of Palm Beach, Loxahatchee Groves, Florida
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Pediatric Neurology PA, Orlando, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Consultants In Epilepsy and Neurology PLLC, Boise, Idaho
  - Carle Foundation Hospital, Urbana, Illinois
  - Midatlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - Mercy Health Saint Mary's Campus, Grand Rapids, Michigan
  - Minnesota Epilepsy Group PA, Saint Paul, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital at Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cincinnati Children's Hospital Medical Center - PIN, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - The University of Pittsburgh, Pittsburgh, Pennsylvania
  - Austin Epilepsy Care Center, Austin, Texas
  - Road Runner Research Ltd, San Antonio, Texas
  - Baylor Scott and White Research Institute, Temple, Texas
  - Clinical Neurosciences Center, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Columbia Saint Mary's, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Wauwatosa, Wisconsin
- Australia (6):
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Austin Health, Heidelberg, Victoria
  - Royal Brisbane & Women's Hospital, Brisbane
  - Royal Melbourne Hospital, Melbourne
  - St Vincent's Hospital Melbourne, Melbourne
  - The Alfred Hospital, Melbourne
- Belgium (5):
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - Hôpital Universitaire des Enfants Reine Fabiola, La Louvière, Hainaut
  - Hôpital Erasme, Brussels
  - UZ Brussel, Jette
  - Centre Neurologique William Lennox, Ottignies-Louvain-la-Neuve
- Czechia (2):
  - Fakultni nemocnice Ostrava, Poruba
  - Thomayerova nemocnice, Prague
- India (9):
  - Synexus Affiliate - Panchshil Hospital, Ahmedabad, Gujarat
  - Synexus Affiliate - Nirmal Hospitals Pvt. Ltd, Surat, Gujarat
  - Synexus Affiliate - Mallikatta Neuro Center, Mangalore, Karnataka
  - Synexus Affiliate - Amrita Institute of Medical Sciences and Research Centre, Kochi, Kerala
  - Synexus Affiliate - Jaslok Hospital and Research Centre, Mumbai, Maharashtra
  - Synexus Affiliate - Kokilaben Dhirubhai Ambani Hospital & Medical Research Institute, Mumbai, Maharashtra
  - Synexus Affiliate - Bharati Hospital, Pune, Maharashtra
  - Nizams Institute of Medical Sciences, Hyderabad
  - Synexus Affiliate - Sir Ganga Ram Hospital, New Delhi
- Japan (8):
  - Eisai Trial Site #1, Fukuoka
  - Eisai Trial Site #3, Fukuoka
  - Eisai Trial Site #7, Hakodate
  - EIsai Trial Site #9, Kagoshima
  - Eisai Trial Site #4, Niigata
  - EIsai Trial Site #8, Osaka
  - Eisai Trial Site #6, Sapporo
  - Eisai Trial Site #2, Shizuoka
- South Korea (4):
  - Kyungpook National University Chilgok hospital, Daegu
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Brigo F, Jones K, Eltze C, Matricardi S. Anti-seizure medications for Lennox-Gastaut syndrome. Cochrane Database Syst Rev. 2021 Apr 7;4(4):CD003277. doi: 10.1002/14651858.CD003277.pub4. PMID 33825230

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 40 investigative sites in Australia, Belgium, the Czech Republic, Japan, India, South Korea, and the United States from 13 December 2016 to 19 July 2021. A total of 101 participants were enrolled (signed informed consent) and 70 participants were randomized to receive study treatment in Core Study Phase.
Pre-assignment Details: This study included a Core Study Phase and an Extension Phase, which in turn consisted of Extension A and Extension B. Study was terminated early by the sponsor due to recruitment challenges that were further impacted by the COVID-19 pandemic.
Groups:
- Core Study Phase: Placebo: Participants received placebo matched to perampanel oral tablets or placebo matched to perampanel oral suspension, once daily at bedtime during the titration period. During the maintenance period, participants continued to receive the placebo matched to perampanel tablets or placebo matched to perampanel oral suspension at dose level that was administered at the end of the titration period. The total duration of the titration period (6 weeks) and maintenance period (12 weeks) in Core Study Phase was 18 weeks.
- Core Study Phase: Perampanel: Participants received starting dose of perampanel, one 2 milligram (mg) oral tablet or 4 milliliter (mL) oral suspension (containing 2 mg perampanel), once daily at bedtime then up-titrated weekly in 2 mg increments to a target dose of 8 milligram per day (mg/day) during titration period. During the maintenance period, participants continued to receive the perampanel dose level that was administered at the end of the titration period. The total duration of the titration period (6 weeks) and maintenance period (12 weeks) in the Core Study Phase was 18 weeks.
- Extension Phase A: Perampanel: Participants who completed the Core Study Phase and who were eligible entered into Extension Phase A. Participants previously assigned to perampanel arm (Core Study Phase) continued taking study medication at the dose received during the Core maintenance period, and participants previously assigned to a placebo arm (Core Study Phase) started perampanel dose as one 2 mg tablet or 4 mL oral suspension (containing 2 mg perampanel) once daily at bedtime, then up-titrated weekly in 2-mg increments up to a maximum dose of 8 mg/day for 6 weeks conversion period of Extension Phase A. After the conversion period, participants could be titrated up to 12 mg/day in 2-week intervals during the maintenance period (46 weeks) of Extension Phase A as per the investigator's discretion. The total duration of the conversion period and maintenance period in Extension Phase A was 52 weeks.
- Extension Phase B: Perampanel: Participants who completed Extension Phase A and who were eligible entered into Extension Phase B. Participants received perampanel at their optimal perampanel dose (that is, dose maintained at the end of Extension A) until perampanel was available commercially or accessible via extended access program (EAP) (in the country in which a participant resides) or unless study termination by the sponsor (up to 188 weeks).
Period: Core Study (Up to 18 Weeks)
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel | Extension Phase A: Perampanel | Extension Phase B: Perampanel
Started | 36 | 34 | 0 | 0
Completed | 32 | 29 | 0 | 0
Not Completed | 4 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 1 | 0 | 0
Period: Extension Phase A (up to 52 Weeks)
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel | Extension Phase A: Perampanel | Extension Phase B: Perampanel
Started | 0 | 0 | 58 (Only eligible participants who completed Core Study entered into Extension Phase A.) | 0
Completed | 0 | 0 | 32 | 0
Not Completed | 0 | 0 | 26 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 0
Not completed — Lack of Efficacy | 0 | 0 | 4 | 0
Not completed — Adverse Event | 0 | 0 | 5 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 9 | 0
Not completed — Other | 0 | 0 | 1 | 0
Period: Extension Phase B (up to 188 Weeks)
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel | Extension Phase A: Perampanel | Extension Phase B: Perampanel
Started | 0 | 0 | 0 | 13 (Only eligible participants who completed Extension Phase A entered into Extension Phase B.)
Completed | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 12
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 8
Not completed — Other | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) was the group of participants who received at least one dose of study drug and had at least one post-dose safety assessment.
Groups:
- Core Study Phase: Perampanel: Participants received starting dose of perampanel, one 2 mg oral tablet or 4 mL oral suspension (containing 2 mg perampanel), once daily at bedtime then up-titrated weekly in 2 mg increments to a target dose of 8 mg/day during titration period. During the maintenance period, participants continued to receive the perampanel dose level that was administered at the end of the titration period. The total duration of the titration period (6 weeks) and maintenance period (12 weeks) in the Core Study Phase was 18 weeks.
- Total: Total of all reporting groups
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (7.80) | 14.7 (10.37) | 14.0 (9.10)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 19 | 16 | 35
  Adolescents (12-17 years) | 7 | 6 | 13
  Adults (18-64 years) | 10 | 12 | 22
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 23 | 17 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 31 | 30 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 13 | 26
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 2 | 6
  White | 15 | 16 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Core Study Phase: Median Percent Change in Drop Seizure Frequency Per 28 Days During Double-blind Treatment Relative to the Prerandomization Phase (Baseline)
Description: Drop seizure was defined as a drop attack or spell involving the entire body, trunk, or head that led to a fall, injury, slumping in a chair, or the participant's head hitting a surface or that could have led to a fall or injury, depending on the participant's position at the time of the attack or spell. Seizure frequency was based on the number of drop seizures per 28 days, calculated as the number of drop seizures over the entire time interval divided by the number of days in the interval and multiplied by 28.
Time Frame: Baseline up to 18 weeks
Population: The full analysis set (FAS) was the group of randomized participants who received at least one dose of the study drug and had at least one post-dose seizure measurement.
Measure: Median (Full Range); unit: percent change
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel
Number analyzed (Participants) | 36 | 34
percent change | -4.51 [-86.2 to 201.8] | -23.07 [-96.4 to 371.4]
Statistical Analysis 1: Comparison: Core Study Phase: Placebo vs Core Study Phase: Perampanel; Test type: Superiority; p = 0.107, ANCOVA — The p-value was based on a rank analysis of covariance (ANCOVA) with treatment, region, and age-group as factors, and prerandomization drop seizure frequency as a covariate; Median Difference (Net) = -19.3, 95% CI 2-sided [-49.2 to 4.8] — The median difference to placebo and the 95 percent (%) confidence interval (CI) were based on the Hodges-Lehmann method

2. Secondary Outcome: Core Study Phase: Median Percent Change in Total Seizure Frequency Per 28 Days During Double-blind Treatment Relative to the Prerandomization Phase (Baseline)
Description: Total seizure was the number of seizures assessed and recorded by the participant's parent/caregiver in the participant seizure diary. Seizure diaries were used to collect seizure counts and types. Seizure frequency was based on the number of drop seizures per 28 days, calculated as the number of drop seizures over the entire time interval divided by the number of days in the interval and multiplied by 28.
Time Frame: Baseline up to 18 weeks
Population: The FAS was the group of randomized participants who received at least one dose of the study drug and had at least one post-dose seizure measurement.
Measure: Median (Full Range); unit: percent change
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel
Number analyzed (Participants) | 36 | 34
percent change | -6.53 [-63.6 to 266.8] | -18.23 [-96.9 to 103.5]

3. Secondary Outcome: Core Study Phase: Percentage of Participants With 50% Response in the Maintenance Period of the Double-blind Treatment Phase Relative to the Prerandomization Phase (Baseline) for Drop Seizures
Description: Drop seizure was defined as a drop attack or spell involving the entire body, trunk, or head that led to a fall, injury, slumping in a chair, or the participant's head hitting a surface or that could have led to a fall or injury, depending on the participant's position at the time of the attack or spell. A responder was a participant who experienced a 50% or greater reduction in drop seizure frequency per 28 days during Maintenance from prerandomization.
Time Frame: Baseline up to 18 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel
Number analyzed (Participants) | 36 | 34
percentage of participants | 25.0 | 44.1

4. Secondary Outcome: Core Study Phase: Percentage of Participants With 50% Response in the Maintenance Period of the Double-blind Treatment Phase Relative to the Prerandomization Phase (Baseline) for Total Seizures
Description: Total seizure was the number of seizures assessed and recorded by the participant's parent/caregiver in the participant seizure diary. Seizure diaries was used to collect seizure counts and types. A responder was a participant who experienced a 50% or greater reduction in drop seizure frequency per 28 days during Maintenance from prerandomization.
Time Frame: Baseline up to 18 weeks
Population: The FAS was the group of randomized participants who received at least one dose of study drug and had at least one post-dose seizure measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel
Number analyzed (Participants) | 36 | 34
percentage of participants | 16.7 | 32.4

5. Secondary Outcome: Core Study Phase: Median Percent Change in Non-drop Seizure Frequency Per 28 Days During Double-blind Treatment Phase Relative to the Prerandomization Phase (Baseline)
Description: Non-drop seizures were defined as non-drop attacks or spells. Drop attacks and spells involved the entire body, trunk, or head and lead to a fall, injury, slumping in a chair, or the participant's head hitting a surface, or could lead to a fall or injury, depending on the participant's position at the time of the attack or spell. Seizure frequency was based on the number of drop seizures per 28 days, calculated as the number of drop seizures over the entire time interval divided by the number of days in the interval and multiplied by 28.
Time Frame: Baseline up to 18 weeks
Population: The FAS was the group of randomized participants who received at least one dose of study drug and had at least one post-dose seizure measurement. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: percent change
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel
Number analyzed (Participants) | 30 | 27
percent change | -13.21 [-100.0 to 2288.1] | -12.33 [-98.7 to 63.2]

6. Secondary Outcome: Core Study Phase: Percentage of Participants With 75% Response in the Maintenance Period of the Double-blind Treatment Phase Relative to the Prerandomization Phase (Baseline) for Drop Seizures, Non-drop Seizures and Total Seizures
Description: Drop seizure was defined as a drop attack or spell involving the entire body, trunk, or head that led to a fall, injury, slumping in a chair, or the participant's head hitting a surface or that could have led to a fall or injury, depending on the participant's position at the time of the attack or spell. Non-drop seizures were defined as non-drop attacks or spells. Total seizure was the number of seizures assessed and recorded by the participant's parent/caregiver in the participant seizure diary. Seizure diaries were used to collect seizure counts and types. A responder was a participant who experienced a 75% or greater reduction in drop seizure/non-drop seizure/ frequency per 28 days during Maintenance from prerandomization.
Time Frame: Baseline up to 18 weeks
Population: The FAS was the group of randomized participants who received at least one dose of the study drug and had at least one post-dose seizure measurement. Here "number analyzed" were participants who were evaluable for the outcome measure at given categories.
Measure: Number; unit: percentage of participants
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel
Number analyzed (Participants) | 36 | 34
percentage of participants
  Drop Seizures | 13.9 | 26.5
  Non-drop Seizures: number analyzed (Participants) | 30 | 27
  Non-drop Seizures | 10.0 | 18.5
  Total Seizures | 0 | 11.8

7. Secondary Outcome: Core Study Phase: Percentage of Participants With 100% Response in the Maintenance Period of the Double-blind Treatment Phase Relative to the Prerandomization Phase (Baseline) for Drop Seizures, Non-drop Seizures and Total Seizures
Description: Drop seizure was defined as a drop attack or spell involving the entire body, trunk, or head that led to a fall, injury, slumping in a chair, or the participant's head hitting a surface or that could have led to a fall or injury, depending on the participant's position at the time of the attack or spell. Non-drop seizures were defined as non-drop attacks or spells. Total seizure was the number of seizures assessed and recorded by the participant's parent/caregiver in the participant seizure diary. Seizure diaries was used to collect seizure counts and types. A responder was a participant who experienced a 100% or greater reduction in drop seizure/non-drop seizure/ frequency per 28 days during Maintenance from prerandomization.
Time Frame: Baseline up to 18 weeks
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel
Number analyzed (Participants) | 36 | 34
percentage of participants
  Drop Seizure | 0 | 2.9
  Non-drop Seizure: number analyzed (Participants) | 31 | 28
  Non-drop Seizure | 6.5 | 3.6
  Total Seizures | 0 | 2.9

8. Secondary Outcome: Core Study Phase: Percentage of Participants With 50% Response in the Maintenance Period of the Double-blind Treatment Phase Relative to the Prerandomization Phase (Baseline) for Non-drop Seizures
Description: Non-drop seizures were defined as non-drop attacks or spells. Drop attacks and spells involved the entire body, trunk, or head and lead to a fall, injury, slumping in a chair, or the participant's head hitting a surface, or could lead to a fall or injury, depending on the participant's position at the time of the attack or spell. A responder was a participant who experienced a 50% or greater reduction in non-drop seizure frequency per 28 days during Maintenance from prerandomization.
Time Frame: Baseline up to 18 weeks
Population: The FAS was the group of randomized participants who received at least one dose of the study drug and had at least one post-dose seizure measurement. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel
Number analyzed (Participants) | 30 | 27
percentage of participants | 16.7 | 44.4

9. Secondary Outcome: Core Study Phase: Percentage of Participants With Clinical Global Impression of Change Scores (CGIC) in the Double-blind Treatment Phase
Description: Assessment of disease severity utilized the CGIC scale at end of treatment to evaluate participants change in disease status from baseline. The CGIC is a 7-point likert scale that measures a physician's global impression of a participants clinical condition. Scale ranged from 1 to 7 with lower score indicated improvement (1=very much improved, 2=much improved, 3=minimally improved), higher score indicated worsening (5=minimally worse, 6= much worse, 7=very much worse), and a score of 4 indicated no change.
Time Frame: Baseline up to 18 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel
Number analyzed (Participants) | 35 | 32
percentage of participants
  Very much improved | 0 | 9.4
  Much improved | 8.6 | 15.6
  Minimally improved | 25.7 | 18.8
  No change | 57.1 | 34.4
  Minimally worse | 5.7 | 12.5
  Much worse | 2.9 | 9.4
  Very much worse | 0 | 0

10. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as an adverse event with an onset date, or a worsening in severity from baseline (pre-treatment), on or after the first dose of study drug up to 28 days following study drug discontinuation. An AE was defined as any untoward medical occurrence in a participant or clinical investigation in a participant administered an investigational product. An AE does not necessarily have a causal relationship with a medicinal product. A serious adverse event (SAE) was defined as any AE if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect.
Time Frame: From the date of the first administration of the study drug up to 28 days after the last dose of the study drug (up to 192 weeks)
Population: SAS was group of participants who received at least one dose of study drug and had at least one post-dose safety assessment. As per the planned safety analysis, safety data for Extension A and Extension B was reported together as 'Extension Phase' arm.
Measure: Count of Participants; unit: Participants
Groups:
- Extension Phase: Perampanel: Participants who completed Core Study and who were eligible entered Extension A. Participants who received perampanel in Core Study, continued at dose received during Core maintenance period, and participants who received placebo in Core Study started perampanel dose as one 2 mg oral tablet or 4 mL oral suspension (containing 2 mg perampanel) once daily at bedtime, then up-titrated weekly in 2-mg increments up to dose of 8 mg/day for 6 weeks conversion period. After conversion period, participants could be titrated up to 12 mg/day in 2-week intervals during maintenance period (46 weeks) as per investigator's discretion. Total duration of conversion and maintenance period in Extension Phase A was 52 weeks. Participants who completed Extension A and who were eligible entered into Extension B in countries where extended access program (EAP) could not be implemented, and received perampanel at optimal dose (dose at end of Extension A) until perampanel was available commercially or unless study termination (up to 188 weeks).
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel | Extension Phase: Perampanel
Number analyzed (Participants) | 36 | 34 | 58
Participants
  TEAEs | 26 | 29 | 50
  SAEs | 1 | 6 | 11

11. Secondary Outcome: Number of Participants With Treatment-emergent Markedly Abnormal Laboratory Values
Description: Treatment-emergent markedly abnormal value for laboratory values was based Common Terminology Criteria for Adverse events (CTCAE) Version 4.0, and determined as if the post baseline CTCAE Version 4.0 grade increases from baseline and the post baseline grade was >=2 (>=3 for phosphate). Laboratory tests included: Hematology count with differential, Chemistry (Electrolytes, Liver function tests, Renal function parameters, Other: albumin, calcium, cholesterol, globulin, glucose, lactate dehydrogenase, phosphorus, total protein, lipid panel, uric acid), Urinalysis, and Viral tests (Hepatitis B surface antigen, Hepatitis C).
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel | Extension Phase: Perampanel
Number analyzed (Participants) | 36 | 34 | 58
Participants
  Markedly Abnormal Low: Platelets | 1 | 0 | 0
  Markedly Abnormal Low: Neutrophils | 0 | 1 | 7
  Markedly Abnormal High: Gamma Glutamyl Transferase | 1 | 1 | 2
  Markedly Abnormal Low: Bicarbonate | 0 | 1 | 1
  Markedly Abnormal High: Sodium | 0 | 1 | 1
  Markedly Abnormal Low: Albumin | 0 | 1 | 0
  Markedly Abnormal High: Cholesterol | 0 | 1 | 1
  Markedly Abnormal High: Triglycerides | 2 | 1 | 4
  Markedly Abnormal Low: Haemoglobin | 0 | 0 | 1
  Markedly Abnormal Low: Lymphocytes | 0 | 0 | 2
  Markedly Abnormal Low: Leukocytes | 0 | 0 | 1
  Markedly Abnormal High: Alanine Aminotransferase | 0 | 0 | 1
  Markedly Abnormal Low: Glucose | 0 | 0 | 1
  Markedly Abnormal High: Alkaline Phosphatase | 0 | 0 | 1

12. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Clinically significant means that a value must have met both the criterion value and satisfied the magnitude of change relative to baseline. Vital sign parameters included systolic blood pressure (BP), diastolic BP, pulse rate.
Time Frame: as for outcome 10
Population: SAS was group of participants who received at least one dose of the study drug and had at least one post-dose safety assessment. As per the planned safety analysis, safety data for Extension A and Extension B was reported together as 'Extension Phase' arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel | Extension Phase: Perampanel
Number analyzed (Participants) | 36 | 34 | 58
Participants
  Systolic Blood Pressure: Low | 4 | 2 | 7
  Systolic Blood Pressure: High | 0 | 0 | 0
  Diastolic Blood Pressure: Low | 5 | 1 | 13
  Diastolic Blood Pressure: High | 0 | 0 | 0
  Pulse Rate: Low | 1 | 0 | 2
  Pulse Rate: High | 4 | 5 | 11

13. Secondary Outcome: Core Study Phase: Model Predicted Average Perampanel Concentrations at Steady State (Cav,ss) During the Maintenance Period of Core Study Phase
Description: Due to the early termination of the study resulting in reduced sample size and the variability in treatment response, population pharmacokinetic (PK) analysis and population pharmacokinetic/pharmacodynamic (PK/PD) modeling planned for this study were not conducted and hence data was not collected and analyzed for this outcome measure.
Time Frame: Up to Week 18
Population: The PK analysis set was the group of participants who received perampanel or placebo who had seizure frequency data with documented dosing history. As population PK and PK/PD analysis were not conducted, therefore data was not collected and analyzed.
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of first administration of study drug up to 28 days after last dose of study drug (up to 192 weeks)
Description: Participants received varying doses in Extension Phase depending on tolerance. Participants were titrated up to 12 mg/day, hence AEs were summarized as a single arm for Extension Phase. As per the planned safety analysis of Extension Phase, safety data for Extension A and Extension B was reported together in a single arm of Extension Phase.
Groups:
- Extension Phase: Perampanel: Participants who completed Core Study and who were eligible entered Extension A. Participants who received perampanel in Core Study, continued at dose received during Core maintenance period; and participants who received placebo in Core Study started perampanel dose as one 2 mg oral tablet or 4 mL oral suspension (containing 2 mg perampanel) once daily at bedtime, then up-titrated weekly in 2-mg increments up to dose of 8 mg/day for 6 weeks conversion period. After conversion period, participants could be titrated up to 12 mg/day in 2-week intervals during maintenance period (46 weeks) as per investigator's discretion. Total duration of conversion and maintenance period in Extension Phase A was 52 weeks. Participants who completed Extension A and who were eligible entered into Extension B in countries where extended access program (EAP) could not be implemented, and received perampanel at optimal dose (dose at end of Extension A) until perampanel was available commercially or unless study termination (up to 188 weeks).
Arm/Group | Core Study Phase: Placebo | Core Study Phase: Perampanel | Extension Phase: Perampanel
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34 | 2/58
Serious Adverse Events (participants affected / at risk) | 1/36 | 6/34 | 11/58
Other Adverse Events (participants affected / at risk) | 26/36 | 29/34 | 50/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Study Phase: Placebo (N=36) | Core Study Phase: Perampanel (N=34) | Extension Phase: Perampanel (N=58)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cytogenetic abnormality (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden unexplained death in epilepsy (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Quadriplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure cluster (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Study Phase: Placebo (N=36) | Core Study Phase: Perampanel (N=34) | Extension Phase: Perampanel (N=58)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Hordeolum (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 2 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (4) | 7 (15)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (7) | 7 (11)
Skin laceration (Injury, poisoning and procedural complications) | 1 (3) | 2 (2) | 3 (4)
Weight increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 6 (6)
Balance disorder (Nervous system disorders) | 0 (0) | 3 (3) | 5 (5)
Drooling (Nervous system disorders) | 1 (1) | 3 (4) | 5 (5)
Lethargy (Nervous system disorders) | 0 (0) | 2 (3) | 2 (3)
Sedation (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2) | 8 (8) | 11 (12)
Agitation (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3)
Irritability (Psychiatric disorders) | 1 (1) | 5 (5) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 4 (4)
Fatigue (General disorders) | 1 (1) | 3 (3) | 4 (4)
Gait disturbance (General disorders) | 0 (0) | 3 (3) | 4 (6)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 5 (5) | 1 (1) | 8 (9)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Study was terminated early by sponsor due to recruitment challenge, further impacted by COVID19, resulting in reduced sample size and variability in treatment response. Population PK analysis and PK/PD modeling planned for this study were not conducted and hence data was not collected and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT02834793/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT02834793/SAP_001.pdf